CLINICAL TRIAL: NCT00963066
Title: NAV-ALI: Effects of Different Levels of Neurally Adjusted Ventilatory Assist (NAVA) in Patients Recovering Spontaneous Breathing After Acute Lung Injury: A Physiological Evaluation.
Brief Title: NAV-ALI: Neurally Adjusted Ventilatory Assist in Patients Recovering Spontaneous Breathing After Acute Lung Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: TERZI Nicolas, CHU de CAEN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-A00583-54
Record Dates: First submitted 2009-08-12; First posted 2009-08-21 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Acute Lung Injury; Mechanical Ventilation
Keywords: NAVA; Acute Lung Injury; Pressure Support Ventilation; Intubation; Tracheostomy; Mechanical ventilation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pressure Support ventilation (Active Comparator)
  Interventions: Device: PSV - pressure suppot ventilation
- NAVA flow triggering (Experimental): Spontaneous Breathing using Neurally Adjusted Ventilatory Assist with flow triggering
  Interventions: Device: NAVA - Neurally Adjusted Ventilatory Assist
- NAVA EMG triggering (Experimental): Spontaneous Breathing using Neurally Adjusted Ventilatory Assist with trigger adjusted on diaphragmatic electromyogram
  Interventions: Device: NAVA - EMG

INTERVENTIONS:
Device: PSV - pressure suppot ventilation — Gold standard partial ventilator support: Pressure Support Ventilation performed with Servo-i® ventilator (MAQUET,Critical Care, Sweden). Different levels of pressure support ventilator assistance are tested.
  Other Names: PSV
  Arms: Pressure Support ventilation
Device: NAVA - Neurally Adjusted Ventilatory Assist — Partial ventilator support with new partial ventilation mode (NAVA) performed with Servo-i® ventilator (Maquet,Critical Care, Sweden). Different levels of neurally adjusted ventilatory assist are tested. Positive pressure, delivered by the machine, is driven using inspiratory flow trigger.
  Other Names: NAVA - Flow
  Arms: NAVA flow triggering
Device: NAVA - EMG — Partial ventilator support with new partial ventilation mode (NAVA) performed with Servo-i® ventilator (Maquet,Critical Care, Sweden). Different levels of neurally adjusted ventilatory assist are tested. The machine applies positive pressure throughout inspiration in proportion to the electrical activity of the diaphragm (Eadi). Eadi was obtained trhough a naso-gastric tube with multiple array of electrodes placed at its distal end (Eadi catheter® , Maquet Critical Care, Sweden).
  Arms: NAVA EMG triggering

SUMMARY:
Evaluation of a new ventilatory mode Neurally Adjusted Ventilatory Assist "NAVA" in patients who recover spontaneous breathing after acute lung injury.

DETAILED DESCRIPTION:
Physiological evaluation of two modes of mechanical ventilation: Neurally Adjusted Ventilatory Assist (NAVA) vs Pressure Support Ventilation, at different levels of ventilator assistance.

Evaluation in term of physiological parameters: Tidal volume, Respiratory rate, Inspiratory effort, PaCO2, evaluation of subject-ventilator synchrony.

Evaluation of physiological response to varying levels of ventilator assistance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hospitalized in intensive care unit
* Acute Lung Injury
* Intubated or tracheotomized and mechanically ventilated

Exclusion Criteria:

* Hemodynamic instability
* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Comparison of physiologic response to varying levels of pressure support and Neurally Adjusted Ventilatory Assist (NAVA) | 24 hours

SECONDARY OUTCOMES:
Subject-ventilator synchrony | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas TERZI, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU de CAEN, Caen, France